CLINICAL TRIAL: NCT06088173
Title: The Effects of Graded Motor Imagery Training Before and After the Rehabilitation Program in Patients With Flexor Tendon Repair
Brief Title: The Effects of Graded Motor Imagery Training Program in Patients With Flexor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, seher karaçam, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUCSD
Record Dates: First submitted 2023-10-08; First posted 2023-10-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Flexor Tendon Repair
Keywords: flexor tendon; Kleinert protocol; graded motor imagery training
MeSH Terms: interventions — Exercise; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Passive Mobilization Group (Experimental): This group will be given Modifiye Kleinert Protocol based rehabilitation
  Interventions: Other: exercises
- Graded Motor Imagery Training Group (Experimental): This group will be given Modifiye Kleinert Protocol and Graded Motor Imagery Training
  Interventions: Other: Exercises and Education

INTERVENTIONS:
Other: exercises — Patients in both group will use Kleinert splint. Sessions will start with ice application if there is edema and continue with scar tissue massage. After general hand massage, passive flexion, active extension exercises; tenodesis exercise and passive punch will be performed for the postoperative (postop) first two weeks. In postop 3-4 weeks, four finger sliding exercises, active half fist and NMES (Neuromuscular electrical stimulation) will be performed. In postop 5-6 weeks, blocking exercises, full punch, grappling hooks and small on-digits holding and releasing exercises will be performed additionally.
  Arms: Early Passive Mobilization Group
Other: Exercises and Education — In addition to the same treatment as the patients in the first group, in the first postoperative (postop) two weeks, the gmi will be explained to the patients and lateralization will be started. lateralization refers to right-left discrimination and the patients will be presented with visuals with the help of the noi recognise app and they will have to decide whether the visual is right or left hand. In the postop 3-4th weeks, the motor imagery stage will be started and imagery will be practiced with the help of the same app. In postop 5-6 weeks, mirror therapy will be practiced with the help of a mirror box.
  Arms: Graded Motor Imagery Training Group

SUMMARY:
The aim of our study was to investigate the effects of graded motor imagery training applied during the immobilization period on hand functions, range of motion, proprioception and kinesiophobia before and after the rehabilitation program in patients with flexor tendon repair.

DETAILED DESCRIPTION:
After flexor tendon repair, conditions such as limitation of joint movement in the injured finger, contracture, decreased proprioception, decreased hand function and skills during activities of daily living may occur due to one or more reasons. Various protocols have been applied in rehabilitation after flexor tendon repair, but the search for new treatment methods to achieve the best results continues. In this study, our aim is to reorganize the cortex and incorporate graded motor imagery training, which has been proven to be more effective in the treatment of chronic pain but promising in terms of increasing body awareness, proprioception and function, into flexor tendon rehabilitation to provide flexor tendon repair patients with more functional results and to contribute to the search for new treatment methods in the literature.

The participants who volunteered to take part in the study will be randomly divided into two groups, namely the Early passive mobilization group (Group 1) and the graded motor imagery (GMI) training (Group 2) using a computerassisted randomization program. After the groups are assigned, Group 1 will receive Modified Kleinert protocol and Group 2 will receive GMI training in addition to Modified Kleinert protocol with the help of hand recognize mobile application. A total of 6 weeks of treatment will be applied. GMI will be taught in sessions and practice will be continued at home. Both groups will use a short modified Kleinert splint for postoperatif 6 weeks. This splint does not allow the use of the hand but allows passive flexion and active extension with the help of a tire. GMI training will be given and practiced as soon as rehabilitation starts. The progression will be 2 weeks lateralization 2 weeks imagery 2 weeks mirror therapy and when the splint is removed at the end of postop 6 weeks. In the remaining sessions, standard rehabilitation will be continued in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Becoming a volunteer
* Being between the ages of 18-65
* Having undergone primary flexor tendon repair
* Being in postoperative week 0-3
* Injury at zone 1-3 level
* At least one of the FDS and FDP tendons is severed
* Be able to use an Android phone

Exclusion Criteria:

* Tendon transfer
* Orthopedic, neurologic, rheumatologic disease in the related extremity
* Associated fracture or nerve injury (except digital nerve)
* Cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Quick-DASH | baseline, postoperative 6th week, postoperatif 8th week
  The QuickDASH is an abbreviated version of the original DASH outcome measure. In comparison to the original 30 item DASH outcome measure, the QuickDASH only contains 11 items. It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level.
Tampa Scale for Kinesiophobia | baseline, postoperative 6th week, postoperatif 8th week
  TSK is a self-reported questionnaire that quantifies fear of movement, or (re)injury. In its original form, the TSK is a 17 item assessment checklist. [1] It uses a 4-point Likert scale (Strongly Disagree-Disagree-Agree-Strongly Agree) with statements that have been later linked to the model of fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury.
Duruöz Hand Index | baseline, postoperative 6th week, postoperatif 8th week
  18 questions regarding ability to carry out manual tasks. Questions are grouped in five domains: In the kitchen (8), dressing (2), hygiene (2), in the office (2), and other (4).
  The patient is instructed to answer each question in terms of the level of difficulty they experience completing various tasks without help from another person or assistive device. Individual items are scored on a 6-point Likert scale where 0=without difficulty and 5=impossible. The 18 individual scores are summed to obtain a composite score The total score ranges from 0-90 with higher scores indicating poorer hand functioning

SECONDARY OUTCOMES:
Active Range of Motion | baseline, postoperative 6th week, postoperatif 8th week
  measured with a finger goniometer
Passive Range of Motion | baseline, postoperative 6th week, postoperatif 8th week
  measured with a finger goniometer
Visual Analog Scale | baseline, postoperative 6th week, postoperatif 8th week
  The patient marks on the line the point that they feel represents their perception of their current state. 0 represents no pain and 10 represents unbearable pa,n. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.

CONTACTS AND LOCATIONS:
Overall Officials: seher DURSUN, Principal Investigator — Istanbul Cerrahpaşa University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Büyükçekmece, Turkey (Türkiye)